CLINICAL TRIAL: NCT06803706
Title: Metabolomic and Gut Microbial Biomarkers of Smoking Cessation Treatment in Long-term Drug Therapy: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1155/2024
Record Dates: First submitted 2025-01-23; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Substance Use Disorder (SUD); Alcohol Use Disorder (AUD); Nicotine Addiction
Keywords: Metabolomics; Gut microbiome; Substance use disorder; nicotine addiction; smoking cessation
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment As Usual (Active Comparator): Patients in the TAU group receive long-term rehabilitation drug treatment according to the 'community as a treatment'-model
  Interventions: Behavioral: Long-term drug therapy within a therapeutic community
- 6-weeks smoking cessation cognitive-behavioral therapy intervention (Experimental): The "smoke free in 6 weeks" program is a standardized behavioural therapy intervention that takes place once a week for 1.5 hours over 6 weeks and is provided by the Austrian health insurance provider Österreichische Gesundheitskasse (ÖGK).
  Interventions: Behavioral: 6-weeks CBT smoking cessation programme; Behavioral: Long-term drug therapy within a therapeutic community

INTERVENTIONS:
Behavioral: 6-weeks CBT smoking cessation programme — Held in the therapeutic community, the intervention will employ principles of cognitive-behavioural therapy (CBT) coupled with personalized recommendations for nicotine replacement. The Austrian Health Insurance standard for therapy will be guiding the program's content, which is tailored for inpatient clients. Specifically, the following interventions based on CBT techniques will be applied in the weekly group sessions consisting of 10 to 15 participants: Psychoeducation including information on tobacco addiction, health risks, advice on relapse prevention and the handling of craving, motivation building, behavioural observation.
  Arms: 6-weeks smoking cessation cognitive-behavioral therapy intervention
Behavioral: Long-term drug therapy within a therapeutic community — The standard treatment within the 'Grüner Kreis' therapeutic community - which all participants will receive - consists of group therapy (once a week), individual psychotherapy (once a week), counselling by social workers, psychiatric consultations, as well as sport-, art- and work-therapy. Daily life is organized according to principles of therapeutic community-based addiction treatment.

SUMMARY:
Theoretical Framework: Cigarette smoking is the leading preventable cause of death worldwide, with nicotine dependence notably common among individuals with Substance Use Disorders (SUD). Smoking exacerbates both physical and mental health issues, further complicating the treatment of SUD. Current therapeutic approaches for SUD often prove inadequate, indicating a need for new strategies. Recent advancements in metabolomics and gut microbiome research have provided valuable insights into the biological mechanisms underlying addiction.

Objectives: This study aims to investigate the therapeutic potential of smoking cessation for individuals with SUD, using a six-week intervention within a therapeutic community. The research specifically explores the psychobehavioral, metabolic, and gut microbiome domains. It is hypothesized that smoking cessation will improve emotional regulation, self-efficacy, and reduce substance craving, mediated by changes in metabolic and microbiome profiles linked to brain reward systems.

Methods: A randomized controlled trial (N=100) will be conducted, examining outcomes such as clinical relapse rates, microbial and metabolic markers, particularly in choline and folate metabolism. Participants will undergo a six-week smoking cessation intervention, with pre- and post-assessments, compared to a control group receiving treatment as usual. Metabolomic and microbiome analyses will be conducted using blood and stool samples, alongside psychological assessments via questionnaires. Assessments on a behavioural level will take place at a 3-months follow-up.

ELIGIBILITY:
Inclusion Criteria: Informed consent, a diagnosis of a form of substance use disorder (F1x.x) by a licensed psychiatrist according to ICD-10, minimum age of 18 years, sufficient knowledge of the German language, willingness to quit smoking.

-

Exclusion Criteria: lack of consent, age below 18, inability to provide informed consent, acute psychotic symptoms or acute suicidal tendencies, cardiovascular disease, pregnancy or breastfeeding, severe mental or organic illnesses (such as epilepsy, brain tumors, recent major surgery), tumor diseases, dementia (Mini Mental Score <20), severe autoimmune diseases or immunosuppression, acute infections, or acute diarrhea, prior gastrointestinal surgery (except appendectomy), probiotic intake within the last 6 months, or those consuming dietary supplements, probiotics, antibiotics, or prebiotic supplements during the study, prior participation in a smoking cessation programme.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | From enrollment to follow-up 3 months after the end of the 6-weeks treatment period
  Self-efficacy as a psychological variable and will be assessed by the Self-Efficacy Scale (SWE), a self-report instrument for measuring general optimistic self-confidence. It consists of 10 items and measures optimistic competence expectancy, i.e., confidence in solving difficult situations with one's own abilities.
General substance-related craving | From enrollment to follow-up 3 months after the end of the 6-weeks treatment period.
  Substance related craving will be assessed by the MaCS (Mannheim Craving Scale). consists of 12 items and four additional items and is rated on a 5- point Likert scale.
Tobacco dependence | From enrollment to follow-up 3 months after the end of the 6-weeks treatment period.
  Tobacco dependence will be assessed by The Fagerström Test for Cigarette Dependence (formerly Fagerström Test for Nicotine Dependence; FTND). It consists of 6 categorically scaled items that assess the number of smoked cigarettes per day (CPD), compulsive use, and dependence intensity.
Primary Affects | From enrollment to follow-up 3 months after the end of the 6-weeks treatment period.
  Primary Affects, as proposed by Jaak Panksepp will be assessed by the German Version of the Brief Affective Neuroscience Personality Scales including a LUST Scale (BANPS-GL), a self-report questionnaire.
Metabolome | From enrollment to the end of the 6-weeks treatment period.
  Metabolome will be ascertained from blood via state-of-the-art NMR (nuclear magnetic resonance).
Gut microbiome | From enrollment to the end of the 6-weeks treatment period.
  Gut microbiome will be ascertained via 16s-rRNA sequencing from stool.
Smoking behaviour | From enrollment to follow-up 3 months after the end of the 6-weeks treatment period.
  Participants will be asked regarding their daily smoked cigarettes in the last two weeks (interval scaled). A second single item question will be, if participants have been completely abstinent from tobacco smoking in the last two weeks (dichotome).

SECONDARY OUTCOMES:
Psychiatric Symptoms | From enrollment to follow-up 3 months after the end of the 6-weeks treatment period.
  For the evaluation of psychopathology, the ICD-10 Symptom Rating (ISR) questionnaire will be utilized. In accordance with the ICD-10, this self-assessment questionnaire, comprising 30 items, is designed to comprehensively assess the status and severity of mental disturbances. Symptoms of the six symptomatic patterns - depressive, anxiety, obsessive-compulsive, eating disorders, somatoform syndrome, and post-traumatic stress disorder - are assessed.

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medical University Graz, Graz
  - Grüner Kreis Organization Johnsdorf Facility, Johnsdorf Brunn
  - Sigmund Freud Private University Vienna, Vienna

REFERENCES:
- [Background] Fuchshuber J, Schober H, Wohlmuth M, Senra H, Rominger C, Schwerdtfeger A, Unterrainer HF. The effectiveness of a standardized tobacco cessation program on psychophysiological parameters in patients with addiction undergoing long-term rehabilitation: a quasi-experimental pilot study. BMC Med. 2024 May 1;22(1):184. doi: 10.1186/s12916-024-03405-z. PMID 38693570